CLINICAL TRIAL: NCT06773806
Title: LIEN ENTRE EXPOSITION A LA CHLORDECONE ET CANCER DE LA PROSTATE EN MARTINIQUE
Brief Title: CHLORDECONE EXPOSURE AND PROSTATE CANCER IN THE FRENCH REGION OF MARTINIIQUE
Acronym: CHLOECAPA
Status: Not yet recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: LABERCA - Laboratoire d'Etude des Résidus et Contaminants dans les Aliments (Unknown); French National Cancer Institute (Institut National Du Cancer - France) (Unknown); Direction Générale de la Santé, France (Other)
Responsible Party: Sponsor
Other Study IDs: C22-52; 2023-A00160-45 (Other: IDRCB)
Record Dates: First submitted 2024-12-19; First posted 2025-01-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Epidemiology; Case-control study; Prostate cancer; Chlordecone; Pesticides
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect blood samples in order to create a serum bank and a DNA bank :
  * The serum bank for the measurement of environmental persistent organic pollutants (POPs), including chlordecone.
  * The DNA bank for the identification of genetic variants at risk of prostate cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prostate cancer patients: The "prostate cancer patients" group consists of :
  * Adult men under 75 years of age,
  * who are resident in Martinique for at least 6 months
  * who have been newly diagnosed with histologically confirmed prostate cancer in Martinique during a given three-year period in all public and private services caring for prostate cancer patients.
- Controls Group 1: The 1st control group also called "negative biopsy group" consists of :
  * Adult men under 75 years of age,
  * who are resident in Martinique for at least 6 months
  * who have had a negative prostate biopsy following elevated PSA (> 2.5 ng/ml) in all public and private services in Martinique identified via urologists or pathologists, during the same given 3-year period as patients,
  * whose the frequency matched on age (+/- 5 years) versus patients
- Controls Group 2: The second control group, also called "PSA negative group", is composed of :
  * Adult men under 75 years of age,
  * who are residing in Martinique for at least 6 months
  * who have had a PSA test less than or equal to the threshold value of 2.5 ng/ml, during the same 3-year period as the patients, identified by a survey institute.
  * whose frequency is age-matched (+/- 5 years) to patients.
  * with quotas defined on socio-professional category in relation to men of the same age residing in Martinique (based on INSEE data).

SUMMARY:
Prostate cancer is the most common male cancer in industrialized countries, including France, with over 60,000 new cases each year, and represents the third leading cause of cancer-related death in men.

The only known risk factors are age, ethnic origin and family history of prostate cancer. Indeed, there are considerable ethnic disparities in prostate cancer risk, with an incidence rate 60% higher in African-American men than in European-American men (Evans 2008). Similarly, in the French West Indies, where over 90% of the population is of Afro-Caribbean origin, the incidence of prostate cancer is twice as high as in mainland France. In 2015, the annual incidence was 88.5 cases per 100,000 in mainland France (Defossez 2021), while it was 184.1 cases per 100,000 in Guadeloupe, over the period 2008-2013 (Desloumeaux 2017), and 161.1 cases per 100,000 in Martinique, over the period 2005-2014 (Joachim 2019). The incidence rates observed in the French West Indies are of the same order as those observed in Afro-Caribbean populations in the UK and African-American populations in the USA (Ben Schlomo 2008, Evans 2008).

The reasons for these ethnic disparities in incidence are still poorly understood, but the role of genetic factors has been suggested. Indeed, certain genetic polymorphisms have been associated with an increased individual risk of prostate cancer in men of sub-Saharan African origin (Conti 2021; Karunamuni 2021; Marlin 2021). In addition, certain environmental factors (in the broadest sense) such as obesity, chronic inflammation, diet and certain environmental pollutants, including persistent organic pollutants (POPs) such as certain organochlorine pesticides, are also strongly suspected.

Among the suspected organochlorine pesticides is chlordecone, an insecticide used in the French West Indies until 1993, strongly suspected of playing a role in the occurrence of prostate cancer, particularly in the West Indies. Indeed, the Kannari study (Dereumeaux and Saoudi 2018), supported by Santé publique France, assessed the exposure of the West Indian population (Martinique and Guadeloupe) in 2013-2014 to chlordecone and certain organochlorine compounds , measured by serum levels, and quantified the determinants of this impregnation. The results of the study show that 90% of the West Indian population is indeed exposed to chlordecone, and demonstrate that chlordecone is still present in the environment (water and soil) and in food products, despite the cessation of its use in the West Indies in 1993.

To date, only one epidemiological study has explored the link between chlordecone exposure and the occurrence of prostate cancer, the Karuprostate study, a case-control study carried out between 2004 and 2007 in Guadeloupe, including 623 prostate cancer cases and 671 controls (Multigner 2010). Chlordecone exposure was measured by serum levels with an initial detection limit of 0.25 μg/L (Multigner 2010), then improved to 0.06 μg/L (Emmeville 2015). The authors highlighted a significant association between chlordecone exposure and prostate cancer, with a positive dose-response relationship (OR=1.77; 95% CI, 1.21 to 2.58 for the highest tercile). This association was more specifically observed in subjects with a family history of prostate cancer and in men who had lived in a Western country, requiring further investigation. The Karuprostate study also showed that serum levels of dichlorodiphenyldichloroethylene (DDE), the main and most stable metabolite of DDT, were significantly associated with the occurrence of CaP (Emmeville 2015). These results underline the interest of assessing, along with chlordecone, co-exposure to other persistent organic or organochlorine pollutants.

Furthermore, DDE exhibits anti-androgenic effects and has been shown to repress the production of Prostatic-Specific Antigen (PSA) (target gene of the androgen receptor) by human prostate cancer cell lines (Wong 2015). The supposed effect of other organochlorines such as chlordecone on androgen receptors and thus on PSA levels could thus have important repercussions in terms of prostate cancer diagnosis. Individual screening for prostate cancer is based on serum PSA levels, followed in cases of elevated PSA (> 3-4 ng/ml) by multiparametric Magnetic Resonance Imaging (mpMRI). A recent study showed that performing pre-biopsy mpMRI, regardless of PSA level, could lead to more men being diagnosed with clinically significant prostate cancer (Eldred-Evans 2021).

Finally, there is a lack of preclinical studies to investigate the distribution of chlordecone in blood and tissues, as well as the link between chlordecone and markers of prostate cancer aggressiveness.

We therefore propose a case-control study in the general population of Martinique. This study will enable us to understand the nature of the link between chlordecone and prostate cancer.

ELIGIBILITY:
INCLUSION CRITERIA

To take part in this research, participants must meet the following criteria:

Patients/cases :

* All men newly diagnosed with Prostate Cancer in Martinique during a three-year given period in all public and private services caring for patients with Prostate Cancer, identified via multidisciplinary consultation meetings.
* Male adults under 75 years of age
* Resident in Martinique for at least 6 months
* Histologically confirmed (inclusion possible as soon as the result is known by the urologist)
* Affiliated to a social security scheme or equivalent
* Have signed a free and informed consent form

Biopsy-negative" controls (Group 1 controls):

* All men with a negative prostate biopsy following elevated Prostate Specific Antigen (PSA) assay (> 2.5 ng/ml) within a 3-year period in all public and private services in Martinique identified via urologists or pathologists.
* Male adults under 75 years of age
* Resident in Martinique for at least 6 months
* Frequency matched on age (+/- 5 years) to patients
* Affiliated to a social security scheme or equivalent
* Signed free and informed consent

PSA-negative" controls (Group 2 controls):

* All men with a PSA ⩽ 2.5 ng/ml within a 3-year period and less than 3 months identified via a survey institute
* Male adults under 75 years of age
* Resident in Martinique for at least 6 months
* Frequency matched on age (+/- 5 years) against patients
* Frequency matched on socio-professional category against men of the same age in Martinique (INSEE data)

NON INCLUSION CRITERIA

To take part in this research, participants must not meet the following criteria:

* Be subject to a legal protection measure (safeguard of justice, curatorship or guardianship).
* Inability to consent because does not speak French or Creole.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological males, given the research focuses on "prostate cancer".
Study Population: Study participants will be selected from the Martinican male population under the age of 80.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure : Measure of association between chlordecone exposure and the risk of prostate cancer. | The blood sample required for chlordecone measurement and the study questionnaire will be taken for each participant during the single inclusion visit. Analysis of the study outcomes will take place at the end of the 36 months recruitment phase.
  Chlordecone exposure will be measured using several complementary methods, combining serum chlordecone assays, an assessment of chlordecone exposure based on questionnaire data (occupational, residential and dietary), and the use of job-exposure or culture-exposure matrices.

SECONDARY OUTCOMES:
Primary secondary outcome measure : Measurement of the association between exposure to chlordecone and other environmental pollutants and serum Prostate-Specific Antigen levels in cases and controls. | From the blood sampling to the statistical analyses it will take about 36 months.
  The association between chlordecone (and other persistent organic pollutants) and PSA levels will be measured using blood tests for these different pollutants.
Secondary secondary outcome measure : Number of significant cancers and aggressive cancers diagnosed on targeted mpMRI biopsies versus number of significant cancers and aggressive cancers diagnosed by systematic biopsies. | It will take around 36 months from recovery of ISUP clinical data to statistical analysis.
  Significant cancer is defined by an ISUP score of 2 or more, and aggressive cancer by an ISUP score > 3 and/or clinical stage T2c or T3.
Third secondary outcome measure: Distribution of chlordecone in blood, adipose and prostate tissue. Validation of a molecular signature, previously identified in vitro, on the cases' tumour tissues. | It will take around 36 months from blood sampling and recovery of the various prostate tissues to analysis of chlordecone distribution and validation of the molecular signature.
  Chlordecone distribution will be investigated by measuring chlordecone levels in blood, periprostatic adipose tissue and prostate tissue from cases treated by radical prostatectomy. A molecular signature associated with chlordecone exposure will be defined in vitro on prostate cancer cell cultures and organotypic cultures of human prostate cancers. This in vitro identified molecular signature will then be validated on tumor tissue from prostate biopsies of the cases, and compared to chlordecone exposure in these patients.
Fourth secondary outcome measure : Genotyping of genetic variants from blood samples using a genome-identity chip. | It will take at least 36 months from blood sampling to genotyping.
  Genetic polymorphisms associated with an increased risk of prostate cancer will be sought and taken into account in the various analyses.

CONTACTS AND LOCATIONS:
Locations (2):
- Martinique (2):
  - The private clinic "Clinique Saint-Paul", Fort-de-France
  - University Hospital of Martinique (CHUM), Fort-de-France

IPD SHARING:
Plan to Share IPD: Undecided